CLINICAL TRIAL: NCT04655170
Title: Randomized, Parallel-group Trial to Evaluate Feasibility, Safety and Efficacy of Nebulized Long-Acting Bronchodilators (Formoterol and Revefenacin) vs. Short-Acting Bronchodilators (Albuterol and Ipratropium) in Hospitalized Patients With AECOPD
Brief Title: Feasibility, Safety and Efficacy of Nebulized Long-Acting Bronchodilators (Formoterol and Revefenacin) vs. Short-Acting Bronchodilators (Albuterol and Ipratropium) in Hospitalized Patients With AECOPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Collaborators: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Principal Investigator, Rajiv Dhand, MD, Professor and Chair Department of Medicine; Division of Pulmonary Medicine Section of Critical Care Medicine, University of Tennessee Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTGSM 4586
Record Dates: First submitted 2020-10-21; First posted 2020-12-07 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: COPD Exacerbation
MeSH Terms: interventions — revefenacin; Formoterol Fumarate

STUDY DESIGN:
Intervention Model Description: Participating patients with AECOPD will be randomized 1:1 to either a standard bronchodilator protocol with nebulized Albuterol and Ipratropium every 6 hours or nebulized Revefenacin 175 μg once per day and Formoterol 20 μg twice per day. Each patient will have a single randomization number indicating the allocated treatment. The treatment assignments will be generated with the use of a pseudo-random-number generator with stratification for age groups (<50, 50-69, >70) that will be used to ensure balance of these factors in the numbers of subjects assigned to each of the two treatments. The allocation to
  treatment arms will be according to a predetermined computer-generated randomization schedule that will not be disclosed to the clinical investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Revefenacin (YUPELRI) & Formoterol (Perforomist) (Experimental): Revefenacin 175 μg once per day and Formoterol 20 μg twice per day via jet nebulizer for 7 days or until discharge if prior to day 7.
  Interventions: Drug: Revefenacin (YUPELRI) & Formoterol (Perforomist)
- Group 2: Ipratropium Bromide (Atrovent) & Albuterol (Ventolin) as Standard of Care (Active Comparator): Albuterol and Ipratropium every 6 hours nebulized over the 7-day treatment period or until discharge if prior to day 7.
  Interventions: Drug: Albuterol Inhalation Aerosol (short-acting beta-agonists) & Ipratropium Aerosol (short-acting anticholinergic)

INTERVENTIONS:
Drug: Revefenacin (YUPELRI) & Formoterol (Perforomist) — Revefenacin is a Long-acting anticholinergics (LAMAs) and Formoterol is Long-acting bronchodilators, beta-agonists (LABAs).
  Arms: Group 1: Revefenacin (YUPELRI) & Formoterol (Perforomist)
Drug: Albuterol Inhalation Aerosol (short-acting beta-agonists) & Ipratropium Aerosol (short-acting anticholinergic) — Albuterol Inhalation Aerosol (short-acting beta-agonists) & Ipratropium Aerosol (short-acting anticholinergic)
  Arms: Group 2: Ipratropium Bromide (Atrovent) & Albuterol (Ventolin) as Standard of Care

SUMMARY:
The purpose of this study is to assess the feasibility, safety and efficacy of a combination of nebulized Formoterol and Revefenacin among patients hospitalized for AECOPD compared with standard-of-care therapy with nebulized Albuterol and Ipratropium.

DETAILED DESCRIPTION:
A prospective, parallel group, randomized clinical trial in 60 patients hospitalized with the primary diagnosis of AECOPD or acute respiratory failure with a secondary diagnosis of COPD (ICD-10 codes J44.1 and J96 - J96.2 with J44.9).

The plan is to:

Administer standard bronchodilator protocol with nebulized Albuterol and Ipratropium every 6 hours (n=30)

versus

Nebulized Revefenacin 175 μg once per day and Formoterol 20 μg twice per day (n=30) for up to 7 days of treatment. Study medication will be administered by standard jet nebulizers in both groups.

Investigators will:

* Collect the Borg dyspnea scale twice a day during hospitalization
* Record the total doses of bronchodilators per day received by each patient
* Record the number of rescue doses needed per day of hospital stay
* Record the lowest level of FiO2 employed on days 1, 3 and 7 of hospital stay
* Record all adverse events and concurrent medications

Investigators will collect:

Physical Exam (Day 1, 3, 7, or ET) Serum Chemistry (Day 1, 3, 7, or ET) Hematology (Day 1, 3, 7, or ET) Chest X-Ray (Day 1).

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Any Race
3. ≥ 40 years of age
4. Admitted to the hospital with a primary diagnosis of AECOPD or acute respiratory failure with a secondary diagnosis of COPD
5. Able to understand and comply with study procedures
6. Willingness to sign and date an Informed Consent Form

Exclusion Criteria:

1. Patients unable or unwilling to sign an informed consent or cooperate with study procedures
2. Patients who are hypersensitive to Formoterol or Revefenacin
3. Patients who are intubated, have tracheotomy, are receiving mechanical ventilation by mask or artificial airway
4. Patients, in the opinion of the investigators, who are rapidly decompensating and are immediately in need, or will soon need, ventilator support
5. Patients who, per the investigator, have unstable cardiovascular disease (e.g., uncontrolled, hypertension, unstable angina, recent MI (within 12 weeks), ventricular arrhythmia, or decompensated heart failure)
6. Patients with a current diagnosis of lung cancer requiring treatment
7. Patients that test positive for COVID-19
8. Pulmonary diseases other than COPD, or lobar pneumonia
9. Patients with acute psychiatric illness deemed significant by the investigator
10. Patients with a history of glaucoma deemed significant by the investigator
11. History of urinary retention deemed significant by the investigator

12 Women who are pregnant or breast feeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Difference in Borg Dyspnea Scale scores between groups | change from baseline borg dyspnea score at day 3
  This is a scale asks the subject to rate the difficulty of their breathing. It starts at number 0 where breathing is causing no difficulty at all and progresses through to number 10 where breathing difficulty is maximal. This will be recorded prior to dosing twice a day between 7 and 9 am & pm. Scores from Group 1 and Group 2 will be averaged and compared.
Difference in Borg Dyspnea Scale scores between groups | change from baseline borg dyspnea score at day 7
  This is a scale asks the subject to rate the difficulty of their breathing. It starts at number 0 where breathing is causing no difficulty at all and progresses through to number 10 where breathing difficulty is maximal. This will be recorded prior to dosing twice a day between 7 and 9 am & pm. Scores from Group 1 and Group 2 will be averaged and compared.
Difference in Borg Dyspnea Scale scores between groups | change from day 3 borg dyspnea score at day 7
  This is a scale asks the subject to rate the difficulty of their breathing. It starts at number 0 where breathing is causing no difficulty at all and progresses through to number 10 where breathing difficulty is maximal. This will be recorded prior to dosing twice a day between 7 and 9 am & pm. Scores from Group 1 and Group 2 will be averaged and compared.
Difference in the mean total doses of short acting bronchodilators (rescue) used during study participation between each group. | up to 7 days
  Subject in both groups will be allowed to use standard of care rescue short-acting bronchodilators throughout their study participation.
The difference in the lowest level of FiO2 employed at each visit between group 1 and group 2 | at baseline
  The lowest level of FiO2 will be recorded from the subjects EMR record at each visit during study participation and the difference between group 1 and group 2 will be noted.
The difference in the lowest level of FiO2 employed at each visit between group 1 and group 2 | at day 3
  The lowest level of FiO2 will be recorded from the subjects EMR record at each visit during study participation and the difference between group 1 and group 2 will be noted.
The difference in the lowest level of FiO2 employed at each visit between group 1 and group 2 | at day 7
  The lowest level of FiO2 will be recorded from the subjects EMR record at each visit during study participation and the difference between group 1 and group 2 will be noted.
Number of total subjects that had to stop treatment early between groups | Through study completion, up to 7 days
  Total percent of patients that had to switch therapy due to lack of response between each group.
The total number of subjects with Adverse Events, SAE's, ET, and Deaths between groups. | Through study completion, up to 7 days
  Adverse Events, SAE's, ET, and Deaths will be recorder for every subjects in both groups until the end of their study participation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided